CLINICAL TRIAL: NCT00790790
Title: A Phase 2 Study of the Effects of LY545694, an iGluR5 Antagonist, in the Treatment of Subjects With Osteoarthritis Knee Pain
Brief Title: A Study in the Treatment of Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11978; H8C-MC-LQBG(a) (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis Knee Pain
MeSH Terms: interventions — dasolampanel etibutil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to LY545694 placebo were given LY545694 placebo twice daily (BID) oral (po) for 5 weeks.
  Interventions: Drug: Placebo
- LY545694 49 mg (Experimental): Participants randomized to LY545694 49 milligrams (mg) BID po were first administered LY545694 21 mg BID po at Visit 3. After 1 week of dosing, participants were escalated to LY545694 49 mg BID po at Visit 4. Participants who were intolerant of this dose were titrated back down to 21 mg BID po for the remainder of study treatment.
  Interventions: Drug: LY545694 49 mg
- LY545694 105 mg (Experimental): Participants randomized to LY545694 105 mg BID po were first administered LY545694 21 mg BID po at Visit 3. After 1 week of dosing, participants were escalated to LY545694 49 mg BID po at Visit 4. At Visit 5, participants were titrated to the final dose of LY545694 105 mg BID po. Participants who were intolerant of this dose were titrated back down to LY545694 49 mg BID po for the remainder of study treatment.
  Interventions: Drug: LY545694 105 mg

INTERVENTIONS:
Drug: Placebo — LY545694 placebo BID po for 5 weeks
  Arms: Placebo
Drug: LY545694 49 mg — LY545694 49 mg BID po for 5 weeks.
  Arms: LY545694 49 mg
Drug: LY545694 105 mg — LY545694 105 mg BID po for 5 weeks.
  Arms: LY545694 105 mg

SUMMARY:
To gather data on whether a new drug for osteoarthritis knee pain will be safe and have an effect on pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Present with Osteoarthritis (OA) of the knee based on: 1) Knee pain for at least 14 days per month for the last 3 months, 2) Osteophytes (bone spurs), 3) And at least 1 of the following: Over the age of 50, OR morning stiffness in knee for less than 30 minutes, OR crunching sensation as the knee bends back and forth (crepitus).
* Mean score of 4 or greater on the 24-hour average pain score from Visit 2 to Visit 3.
* Completion of electronic daily diaries with at least 70% complete between Visit 2 and Visit 3.
* Taken non-steroidal anti-inflammatory drugs (NSAIDs) less than 15 days over the past month AND not taken NSAIDs at least 1 week prior to Visit 3.
* Agree to maintain the same activity level throughout the study.
* Women who can become pregnant must test negative for pregnancy and agree to utilize medically acceptable/reliable birth control during the study and 1 month following the last dose of the study.
* Competent and freely able to give an informed consent.
* Ability to understanding and intelligibly communicate with the investigator.
* Judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures required by the protocol.

Exclusion Criteria:

* Knee arthroscopy within past 3 months or any knee joint replacement.
* Surgery planned during the trial for the knee to be studied.
* Prior synovial fluid analysis showing a white blood cell of 2000 cubic millimeters (mm^3) that is indicative of a diagnosis other than OA
* Are non-ambulatory or require the use of crutches or a walker. Use of a cane in the hand opposite the index knee is acceptable.
* Body Mass Index over 40.
* Confounding painful condition that may interfere with assessment of the index knee. (Knee pain should be the predominant pain. Mild OA of the hands is allowed, for instance.)
* Diagnosis of inflammatory arthritis (rheumatoid arthritis) or an autoimmune disorder (except inactive Hashimoto's thyroiditis).
* Received intra-articular hyaluronate or steroids, joint lavage, or other invasive therapies to the knee in the past 3 months.
* Frequent falls that could result in hospitalization or could compromise response to treatment.
* Current or previous (within the past 1 year) Axis 1 diagnosis of major depressive disorder, mania, bipolar disorder, psychosis, dysthymia, anxiety disorder, alcohol or eating disorders.
* Serious or unstable cardiovascular, hepatic, renal, respiratory, ophthalmologic, gastrointestinal, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition that in the opinion of investigator would compromise participation or be likely to lead to hospitalization during the course of the study.
* Alanine transaminase (ALT) > 2.0 times upper limit of normal at Visit 1, based on reference ranges of the central lab.
* Prior renal transplant, current renal dialysis, or serum creatinine laboratory value >1.5 times upper limit of normal based on the reference ranges of the central lab.
* Diagnosis or past history of glaucoma. Subjects with intraocular pressure >24 millimeters of mercury (mm Hg).
* Are taking any excluded medications that cannot be discontinued at Visit 1.
* History of substance abuse or dependence within the past year, excluding nicotine and caffeine. Have a positive urine drug screen for any substance of abuse or excluded medication.
* History of recurrent seizures other than febrile seizures.
* Are judged by the investigator to be at suicidal risk.
* History of frequent and/or severe allergic reactions with multiple medications.
* Pregnant or breast-feeding.
* Are unwilling/unable to comply with the use of a data collection devices.
* Received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Investigator site personnel directly affiliated with this study, and/or their immediate families, or Lilly employees.
* History of severe delay in stomach emptying (gastroparesis).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edison, New Jersey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey, Puerto Rico
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period 1 was an up to 5-week screening phase when participants stopped use of excluded medications (265 participants entered; 118 discontinued). Study Period 2 was a 5-week, double-blind therapy period when randomization and dispensing of study drug occurred. Study Period 3 was a 1-week washout phase when all study medication was stopped.
Period: Study Period 2: Therapy Phase
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Started | 49 | 50 | 48
Completed | 37 | 32 | 27
Not Completed | 12 | 18 | 21
Not completed — Adverse Event | 3 | 16 | 16
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 2
Not completed — Lack of Efficacy | 1 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0
Period: Study Period 3: 1-Week Washout Phase
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Started | 37 | 32 | 27
Completed | 37 | 31 | 26
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg | Total
Number analyzed (Participants) | 49 | 50 | 48 | 147
Age Continuous [Mean (Standard Deviation); unit: years] | 59.59 (6.81) | 57.68 (7.88) | 59.96 (6.98) | 59.06 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 33 | 101
  Male | 15 | 16 | 15 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 2 | 0 | 5
  Black or African American | 5 | 6 | 5 | 16
  Multiple | 2 | 0 | 0 | 2
  White | 39 | 42 | 43 | 124
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 31 | 94
  Puerto Rico | 7 | 8 | 8 | 23
  Romania | 11 | 10 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Mean 24-hour Average Pain Severity (APS) Score From Electronic Diary at 5 Weeks
Description: This scale measured 24-hour APS scores. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Least Squares (LS) Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either LY545694 or placebo treatment with both baseline and at least 1 postbaseline measure. Last observation carried forward (LOCF) was conducted on the primary efficacy measure modified ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 32 | 27
units on a scale | -2.05 (0.29) | -2.10 (0.29) | -2.09 (0.30)

2. Secondary Outcome: Change From Baseline in Weekly Mean Night Pain Severity Score From Electronic Diary at 5 Weeks
Description: This scale measured night pain APS scores. Data were recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either LY545694 or placebo treatment with both baseline and at least 1 postbaseline measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 32 | 27
units on a scale | -2.22 (0.31) | -2.13 (0.32) | -2.19 (0.33)

3. Secondary Outcome: Change From Baseline in Weekly Mean Worst Daily Pain Severity Score From Electronic Diary at 5 Weeks
Description: This scale measured worst pain APS scores. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 32 | 27
units on a scale | -2.12 (0.30) | -2.37 (0.31) | -2.09 (0.32)

4. Secondary Outcome: Number of Participants With 30% Reduction in Weekly Mean 24-hour Average Pain Severity (APS) Score
Description: This scale measured 24-hour APS scores. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point Likert scale was also used for assessment of night pain and worst pain each day, evaluated as weekly means.
Time Frame: Baseline through 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either LY545694 or placebo treatment with both baseline and at least 1 postbaseline measure. LOCF was conducted on the primary efficacy measure modified ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 49 | 48 | 47
participants | 17 | 17 | 21

5. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at 5 Weeks
Description: CGI-S measured severity of illness at the time of assessment compared with start of treatment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale | -1.09 (0.16) | -1.04 (0.17) | -1.03 (0.18)

6. Secondary Outcome: Change From Baseline in Average Brief Pain Inventory - Interference (BPI-I) Subscale Score at 5 Weeks
Description: Average BPI-I was a self-reported scale measuring degree of pain interference on function. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessed interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale | -2.12 (0.35) | -2.07 (0.36) | -1.39 (0.38)

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory - Severity (BPI-S) Subscale Score at 5 Weeks
Description: BPI-S was a self-reported scale measuring severity of pain. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessed worst pain, least pain, and average pain in past 24 hours, and current pain. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale
  BPI-S Worst Pain | -2.32 (0.38) | -2.78 (0.40) | -2.48 (0.43)
  BPI-S Least Pain | -1.59 (0.34) | -1.99 (0.34) | -1.84 (0.36)
  BPI-S Average Pain | -1.99 (0.31) | -2.30 (0.32) | -1.91 (0.35)
  BPI-S Current Pain | -2.18 (0.36) | -2.36 (0.37) | -2.09 (0.40)

8. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score at 5 Weeks
Description: PGI-I was a scale that measured the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranged from 1 (very much better) to 7 (very much worse). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale | 2.89 (0.23) | 2.73 (0.24) | 2.96 (0.25)

9. Secondary Outcome: Change From Baseline in Assessment of Sleep Questionnaire (ASQ) Total Score at 5 Weeks
Description: ASQ consisted of 21 items (including a single item to assess overall sleep quality) and 3 subscales: Sleep Onset and Maintenance (items 1-3, 5-6, 9, 11); Sleep Experience (items 4, 7, 8, 10, 12); and Awakening Experience (items 13-20). Each item was scored on a 5-point Likert scale, ranging from 0 (no sleep at all) to 5 (a lot of sleep). Each subscale was calculated as the mean of the individual items comprising the subscale. A total ASQ score was calculated as the mean of the subscale scores; higher scores represented better sleep.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale | 0.24 (0.12) | 0.22 (0.12) | 0.20 (0.13)

10. Secondary Outcome: Change From Baseline in Total Western Ontario and MacMaster (WOMAC) Osteoarthritis Physical Function, Pain, and Stiffness Subscales at 5 Weeks
Description: The Total WOMAC index (pain, stiffness, physical function subscales) was completed by the participant and had 24 questions. Each question was answered using a 5-point Likert scale (0 to 4). The Total score had a range from 0 (none) to 96 (extreme). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
units on a scale | -18.03 (2.83) | -18.44 (2.94) | -19.92 (3.15)

11. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Health Survey Bodily Pain Score at 5 Weeks
Description: The SF-36 Health Status Survey was a generic, health-related scale assessing participants' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicated better health status). Domain scores: general health=5-25; physical functioning=10-30; role-physical=4-8; role-emotional=3-6; social functioning=2-10; bodily pain=2-11; vitality=4-24; mental health=5-30.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 46 | 44 | 41
units on a scale | 1.10 (0.30) | 1.59 (0.30) | 1.24 (0.31)

12. Secondary Outcome: Change From Baseline in European Quality of Life Scale - 5 Dimensions (EQ-5D) at 5 Weeks: United States Population Based Index Score
Description: The EuroQoL Questionnaire - 5 Dimension (EQ-5D) was a generic, multidimensional, health-related, quality-of-life instrument. The profile allowed participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 was generated for each domain. For each participant, the outcome rating on the 5 domains was mapped to a single index through an algorithm. The index ranged between 0 and 1, with the higher score indicating a better health state perceived by the participant.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 47 | 46 | 45
units on a scale | 0.11 (0.03) | 0.07 (0.03) | 0.05 (0.03)

13. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Global Impairment Score at 5 Weeks
Description: The SDS was completed by the participant and was used to assess the effect of the participant's symptoms on their work/social/family life. Total scores ranged from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 46 | 47 | 44
units on a scale | -3.36 (1.08) | -2.73 (1.06) | -2.86 (1.10)

14. Secondary Outcome: Number of Participants Who Discontinued Due to Treatment Emergent Adverse Events (TEAEs) During the Therapy Phase and 1-Week Washout Phase
Description: Participant discontinuation in the study due to serious and other non-serious AEs was measured during both the therapy (double-blind) phase and 1-week washout (follow-up) phase. A listing of serious and other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 6 weeks
Population: The safety analysis population included all 147 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 49 | 50 | 48
participants
  Therapy Phase | 3 | 16 | 16
  1-Week Washout Phase | 0 | 0 | 1

15. Secondary Outcome: Number of Participants With Serious Treatment Emergent Abnormal High or Low Laboratory Values
Description: The number of participants by treatment group who had abnormal high or low laboratory values was summarized as serious adverse events (SAEs) from the "Investigations" system organ class during the treatment phase of the study. A listing of SAEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 5 weeks
Population: The safety analysis population included all 147 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 49 | 50 | 48
participants | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure and Diastolic Blood Pressure at 5 Weeks
Description: Participants' systolic blood pressure and diastolic blood pressure were measured in millimeters of mercury (mmHg). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
millimeters of mercury (mmHg)
  Systolic Blood Pressure (mmHg) | -2.13 (1.81) | -2.50 (1.87) | -2.15 (2.03)
  Diastolic Blood Pressure (mmHg) | -2.00 (1.16) | -0.49 (1.20) | -0.39 (1.30)

17. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate at 5 Weeks
Description: Pulse rate was measured in beats per minute (bpm). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
beats per minute (bpm) | 0.06 (1.13) | 0.59 (1.19) | 2.17 (1.32)

18. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Change in Heart Rate Using Bazett's (QTcB) and Fridericia's (QTcF) Formulas
Description: The number of participants having QTcF and QTcB ECG change >450 milliseconds (msec) was summarized.
Time Frame: Baseline through 5 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 47 | 46 | 43
participants
  QTcB >450 msec | 2 | 2 | 4
  QTcF >450 msec | 1 | 1 | 2

19. Secondary Outcome: Number of Participants Reporting Blurry or Hazy Vision Using the Subjective Vision Inventory (SVI) Question 1 (Q1) at 5 Weeks
Description: This scale first asked if the participant was experiencing hazy or blurry vision or if he/she had difficulty focusing. If the answer was yes, followup questions rated the degree to which the issue impaired his/her ability to do work or read.
Time Frame: Week 5
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 37 | 33 | 27
participants
  Yes | 0 | 1 | 1
  No | 37 | 32 | 26

20. Secondary Outcome: Pharmacokinetic (PK) Parameter: Clearance of LY545694 (CLp) and Compound 645838 (CLm)
Description: Clearance was the volume of plasma cleared of study drug LY545694 (CLp) and metabolite compound 645838 (CLm) per unit time. The original PK/pharmacodynamic (PD) relationship outcome measure analysis was not conducted; therefore, only PK data were reported.
Time Frame: Baseline through 5 weeks
Population: The PK dataset for population modeling consisted of quantifiable plasma LY545694 and Compound 64538 concentrations from participants following daily oral doses of LY545694 21 mg to LY545694 105 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour (L/hr)
Groups:
- LY545694 Clearance (CLp): Plasma LY545694 concentrations were obtained following daily oral doses of LY545694 21 mg to LY545694 105 mg.
- Compound 645838 (CLm): Plasma Compound 645838 concentrations were obtained following daily oral doses of LY545694 21 mg to 105 mg.
Arm/Group | LY545694 Clearance (CLp) | Compound 645838 (CLm)
Number analyzed (Participants) | 91 | 91
Liter per hour (L/hr) | 90.5 [71.8 to 115.0] | 41.9 [37.4 to 47.6]

21. Secondary Outcome: Number of Participants With Neurological Treatment Emergent Adverse Events (AEs)
Description: The total number of TEAEs (serious and non-serious) that first occurred or worsened during the treatment period) from the "Nervous system disorders" system organ class was summarized. A listing of serious and other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 5 weeks
Population: The safety analysis population included all 147 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 49 | 50 | 48
participants | 4 | 14 | 17

22. Secondary Outcome: Time to Response
Description: Time to response=first visit achieving a 30% reduction of weekly mean 24-hour APS score. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The number of days at which 30% of the participants at risk had at least 30% response was reported.
Time Frame: Baseline through 5 weeks
Population: as for outcome 2
Measure: Number; unit: Time (days)
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 49 | 48 | 47
Time (days) | 28 | 16 | 24

ADVERSE EVENTS:
Groups:
- LY545694 49 mg: Participants randomized to LY545694 49 milligrams (mg) twice daily (BID) oral (po) were first administered LY545694 21 mg BID po at Visit 3. After 1 week of dosing, participants were escalated to LY545694 49 mg BID po at Visit 4. Participants who were intolerant of this dose were titrated back down to 21 mg BID po for the remainder of study treatment.
- Placebo Washout: 1 week washout period from taking placebo
- LY545694 49 mg Washout: 1 week washout period from taking 49 mg LY545694
- LY545694 105 mg Washout: 1 week washout period from taking 105 mg LY545694
Arm/Group | Placebo | LY545694 49 mg | LY545694 105 mg | Placebo Washout | LY545694 49 mg Washout | LY545694 105 mg Washout
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/50 | 1/48 | 0/49 | 1/50 | 0/48
Other Adverse Events (participants affected / at risk) | 23/49 | 34/50 | 33/48 | 1/49 | 4/50 | 2/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | LY545694 49 mg (N=50) | LY545694 105 mg (N=48) | Placebo Washout (N=49) | LY545694 49 mg Washout (N=50) | LY545694 105 mg Washout (N=48)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | LY545694 49 mg (N=50) | LY545694 105 mg (N=48) | Placebo Washout (N=49) | LY545694 49 mg Washout (N=50) | LY545694 105 mg Washout (N=48)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Presbyopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 10 (13) | 17 (23) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 6 (8) | 11 (14) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 6 (8) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Expressive language disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition frequency decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Verbal abuse (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days